CLINICAL TRIAL: NCT04221373
Title: The Effects of Incorporated Exoskeletal-Assisted Walking in Spinal Cord Injury (SCI) Acute Inpatient Rehabilitation
Brief Title: Exoskeletal-Assisted Walking in SCI Acute Inpatient Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Ann M. Spungen EdD, Vice Chairperson of Research, Department of Rehabilitation and Human Performance, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 18-1632; DOH01-C34722GG-3450000 (Other Grant/Funding Number: Department of Health, State of New York)
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Spinal Cord Injuries; Inpatient
Keywords: Rehabilitation; Walking; Exoskeletons
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A two-group, single blinded (raters are not part of intervention) and randomized clinical trial (RCT) with stratification for traumatic or non-traumatic injury will be performed. A total of 30 people with non-progressive SCI, who are over 18 years and eligible for locomotor training as part of acute inpatient rehabilitation (AIR) will be randomized. We expect to recruit, consent, and screen 40 people to accommodate a 25% drop-out rate due to unpredictability during inpatient stay for a target sample of 30 participants to complete the protocol. Eligible participants will be randomized into either the intervention group or the control group. Each group will have 15 participants stratified for 7 having traumatic and 8 having non-traumatic etiologies
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors are not part of intervention. They will not know which group participants will be in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Exoskeletal-assisted walking training group (Experimental): Participants will receive locomotor training provided with an Ekso™ powered exoskeleton according to the standard of care of AIR at Mount Sinai Hospital with the exception that the EAW training will be incorporated into the designated therapy times (3 hours of physical therapy (PT) and/or occupational therapy (OT)) which will be provided as determined by the clinical team from the earliest time they are identified to be able to safely stand, through discharge. The goal of EAW intervention is to complete three or more sessions of EAW training a week during the AIR period (after enrolling into the study until discharge).
  Interventions: Device: Ekso™ powered exoskeleton; Other: Standard of care
- Standard of care group (Active Comparator): Participants will receive standard of care of acute inpatient rehabilitation which includes three hours of physical therapy and/or occupational therapy per day until they are discharged.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: Ekso™ powered exoskeleton — Powered exoskeletal-assisted walking (EAW) for early training
  Arms: Exoskeletal-assisted walking training group
Other: Standard of care — Participants will receive standard of care of acute inpatient rehabilitation.

SUMMARY:
The purpose of this research study is to test the effect of early exoskeletal-assisted walking (EAW) training (combined into regular acute inpatient rehabilitation (AIR)) on improving functional recovery and reducing pain and inflammation. Powered exoskeletons are a technology that offer standing and walking for certain persons with spinal cord injury (SCI) who meet the using indication of the device and have been used in the chronic SCI population with positive benefits in ability to move, daily function (such as bathing and dressing), body composition (such as lean and fat tissue mass), and quality of life (QOL). Despite the potential for EAW to promote functional recovery and reduce secondary medical complications (such as urinary tract infections and pain), no reports exist on the use of exoskeletons in AIR.

DETAILED DESCRIPTION:
People with spinal cord injury (SCI) can have an abrupt loss of upright mobility, function and physical activity. Inflammation and pain are reported to be increased, with negative impacts on quality of life. Powered exoskeletons are a technology that offer standing and walking for eligible persons with SCI and have predominantly been used in the chronic SCI population with positive benefits in mobility, function, body composition, and quality of life (QOL). Despite the potential for exoskeletal-assisted walking (EAW) to promote functional recovery and mitigate secondary medical complications, no reports exist on the use of exoskeletons in acute inpatient rehabilitation (AIR). The goal of this study is to test the effect of early EAW training (incorporated into regular AIR) on accelerating functional recovery and reducing pain and inflammation. A total of 30 people with non-progressive SCI (≥18 years; <6 months after SCI), who are clinically eligible for gait training during AIR, will be randomly assigned into one of two groups (15 participants/group, stratified evenly for traumatic and non-traumatic SCI). The intervention group will receive gait training with an Ekso powered exoskeleton, incorporated into usual 3-hour AIR (AIR with EAW group). The control group will have usual 3-hour AIR, but without using an exoskeleton (AIR only group). Motor function, functional activities, pain and inflammation will be assessed after enrollment in the study and before discharge from AIR. The intervention group is expected to have significantly better outcomes compared with the control group. The impact of successful completion of this study would increase knowledge of the effect of using EAW during acute/subacute AIR. The expected outcome of this study is that exoskeletal-assisted walking during AIR will have significantly greater effects on mitigating some of the secondary consequences of paralysis from SCI during the early phases of recovery and rehabilitation.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or greater
* Height between 5'2" and 6'2" (1.6 meters to 1.9 meters)
* Weight less than 220 pounds (100 kilograms)
* Hip: 5 degrees of extension; 110 of flexion
* Knee: Full extension to 110 of flexion
* Ankle: at least 0 of dorsiflexion to 25 of plantarflexion
* Are eligible for locomotor training as part of inpatient rehabilitation
* Independent with static sitting balance
* Sufficient function upper extremity strength to manage walking aid (front-wheeled walker, platform walker, or crutches)
* Able to follow directions

Exclusion Criteria

* Uncontrolled cardiovascular conditions (i.e. heart failure, angina, hypertension)
* Inability to stand upright due to orthostatic hypotension
* Any form of progressive SCI as defined by the physician, such as cancers
* Body characteristics that do not fit within exoskeleton limits
* Upper leg length discrepancy > 0.5" or lower leg discrepancy >0.75"
* Skin integrity issues in areas that would contact the device or that would likely be made worse by device use
* Pregnancy
* Colostomy
* Mechanical ventilation
* Non-English Speaking
* The participant is able to walk better with exoskeleton assistance at baseline
* Any other issue that might prevent safe standing or walking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Spungen, Ed.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kozlowski AJ, Bryce TN, Dijkers MP. Time and Effort Required by Persons with Spinal Cord Injury to Learn to Use a Powered Exoskeleton for Assisted Walking. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):110-21. doi: 10.1310/sci2102-110. Epub 2015 Apr 12. PMID 26364280
- [Background] Yang A, Asselin P, Knezevic S, Kornfeld S, Spungen AM. Assessment of In-Hospital Walking Velocity and Level of Assistance in a Powered Exoskeleton in Persons with Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2015 Spring;21(2):100-9. doi: 10.1310/sci2102-100. Epub 2015 Apr 12. PMID 26364279
- [Background] Bach Baunsgaard C, Vig Nissen U, Katrin Brust A, Frotzler A, Ribeill C, Kalke YB, Leon N, Gomez B, Samuelsson K, Antepohl W, Holmstrom U, Marklund N, Glott T, Opheim A, Benito J, Murillo N, Nachtegaal J, Faber W, Biering-Sorensen F. Gait training after spinal cord injury: safety, feasibility and gait function following 8 weeks of training with the exoskeletons from Ekso Bionics. Spinal Cord. 2018 Feb;56(2):106-116. doi: 10.1038/s41393-017-0013-7. Epub 2017 Nov 6. PMID 29105657
- [Background] Forrest GF, Sisto SA, Barbeau H, Kirshblum SC, Wilen J, Bond Q, Bentson S, Asselin P, Cirnigliaro CM, Harkema S. Neuromotor and musculoskeletal responses to locomotor training for an individual with chronic motor complete AIS-B spinal cord injury. J Spinal Cord Med. 2008;31(5):509-21. doi: 10.1080/10790268.2008.11753646. PMID 19086708
- [Derived] Tsai CY, Weinrauch WJ, Manente N, Huang V, Bryce TN, Spungen AM. Exoskeletal-Assisted Walking During Acute Inpatient Rehabilitation Enhances Recovery for Persons with Spinal Cord Injury-A Pilot Randomized Controlled Trial. J Neurotrauma. 2024 Sep;41(17-18):2089-2100. doi: 10.1089/neu.2023.0667. Epub 2024 May 8. PMID 38661533

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exoskeletal-assisted Walking Training Group | Standard of Care Group
Started | 20 | 12
Completed | 16 | 12
Not Completed | 4 | 0
Not completed — Physician Decision | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exoskeletal-assisted Walking Training Group | Standard of Care Group | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (18.3) | 46.8 (18.3) | 46.3 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Etiology [Count of Participants; unit: Participants]
  traumatic | 13 | 9 | 22
  non-traumatic | 3 | 3 | 6
Neurological Level of Injury (NLI) [Count of Participants; unit: Participants]
  cervical | 7 | 5 | 12
  thoracic | 5 | 4 | 9
  lumbar | 4 | 3 | 7
ASIA Impairment Scale (AIS) [Count of Participants; unit: Participants] — American Spinal Injury Association Impairment Scale (AIS):
  A - Complete Injury - No sensory or motor function
  B - Sensory Incomplete - Sensory but not motor function is preserved below the neurological level
  C- Motor Incomplete - Motor function is preserved below the neurological level
  Participants
    A - Complete | 3 | 4 | 7
    B - Sensory Incomplete | 4 | 2 | 6
    C - Motor Incomplete | 9 | 6 | 15
Inpatient Stay Days [Mean (Standard Deviation); unit: days] | 51.6 (18.7) | 41.8 (21.0) | 47.4 (19.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Spinal Cord Independence Measure (SCIM) Version III Scores
Description: Functional activities will be assessed using Spinal Cord Independence Measure (SCIM) scores evaluated by clinicians. Full Scale range from 0-100, higher score indicates more independence. Each subscale score is evaluated within the 100-point scale (self-care: 0-20; respiration and sphincter (R & S) management: 0-40; mobility: 0-40)
Time Frame: Baseline and before discharge from acute inpatient rehabilitation (average 2-3 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeletal-assisted Walking Training Group | Standard of Care Group
Number analyzed (Participants) | 16 | 12
score on a scale
  Total score, baseline | 18.6 (6.4) | 27.0 (12.3)
  Total score before discharge, 2-3 weeks | 54.5 (13.8) | 50.0 (20.0)
  Self-care subscore, baseline | 5.5 (4.7) | 7.2 (3.9)
  Self-care subscore, before discharge, 2-3 weeks | 14.1 (4.9) | 12.6 (6.9)
  R&S management subscore, baseline | 11.4 (2.7) | 18.2 (8.0)
  R&S management subscore before discharge, 2-3 weeks | 26.3 (6.6) | 25.6 (8.1)
  Mobility subscore, baseline | 1.7 (2.4) | 1.7 (2.9)
  Mobility subscore, before discharge, 2-3 weeks | 14.2 (4.7) | 11.8 (6.9)
Statistical Analysis 1: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; SCIM Total Score; Test type: Other — Mixed-effects model; p < 0.01, Mixed Models Analysis — Main effect of time; F(1, 26) = 117.78
Statistical Analysis 2: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; SCIM Total Score; Test type: Other — Mixed-effects model; p = 0.03, Mixed Models Analysis — treatment group by time interaction effects; F(1,26) = 5.59
Statistical Analysis 3: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; SCIM R & S scores; Test type: Other — Mixed-effects model; p = 0.01, Mixed Models Analysis — treatment group by time interaction effects; F(1,26) = 8.02
Statistical Analysis 4: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; SCIM R & S scores; Test type: Other — Mixed-effects model; p < 0.01, Mixed Models Analysis — Main effect of time; F(1, 26) = 72.49

2. Secondary Outcome: Change in International Standards for Neurological Classification of SCI (ISNCSCI)
Description: Motor and sensory function was assessed by a physiatrist using the International Standards 152 for Neurological Classification of Spinal Cord Injury (ISNCSCI) to determine a total motor score (TMS, ranges from 0 to 100), upper extremity motor score (UEMS, ranges from 0 to 50), lower extremity motor score (LEMS, ranges from 0 to 50), total light touch score (TLTS, ranges from 0 to 112), total pin prick score (TPPS, ranges from 0 to 112), and total sensory score (TSS, ranges from 0 to 224). Higher score indicates better function.
Time Frame: Baseline and before discharge from acute inpatient rehabilitation (average 2-3 weeks)
Population: Some participants had missing data because they rejected conducting the full ISNCSCI sensory test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeletal-assisted Walking Training Group | Standard of Care Group
Number analyzed (Participants) | 16 | 12
score on a scale
  Lower extremity motor score (LEMS), baseline | 8.8 (9.3) | 10.7 (9.8)
  LEMS, before discharge, 2-3 weeks | 24.2 (12.4) | 17.0 (11.6)
  Upper extremity motor score, before discharge, baseline | 35.8 (15.9) | 40.3 (14.6)
  UEMS, before discharge, 2-3 weeks | 42.6 (9.9) | 42.3 (12.4)
  Total Motor Score (TMS), baseline | 44.6 (17.5) | 51.0 (16.5)
  TMS before discharge, 2-3 weeks | 66.8 (13.1) | 59.3 (15.1)
  TLTS, baseline: number analyzed (Participants) | 13 | 10
  TLTS, baseline | 78.5 (15.5) | 80.8 (24.6)
  TLTS, before discharge, 2-3 weeks: number analyzed (Participants) | 13 | 10
  TLTS, before discharge, 2-3 weeks | 90.0 (16.9) | 80.2 (27.6)
  TPPS, baseline: number analyzed (Participants) | 12 | 10
  TPPS, baseline | 70.0 (23.9) | 72.7 (30.1)
  TPPS, before discharge, 2-3 weeks: number analyzed (Participants) | 12 | 10
  TPPS, before discharge, 2-3 weeks | 84.5 (16.6) | 76.3 (30.4)
  TSS, baseline: number analyzed (Participants) | 11 | 9
  TSS, baseline | 144.0 (37.1) | 151.4 (56.1)
  TSS, before discharge, 2-3 weeks: number analyzed (Participants) | 11 | 9
  TSS, before discharge, 2-3 weeks | 170.1 (32.5) | 155.1 (60.4)
Statistical Analysis 1: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; LEMS; Test type: Other — Mixed-effects model; p = 0.02, Mixed Models Analysis — Treatment group by time interaction effects; F(1,26) = 5.82
Statistical Analysis 2: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; LEMS; Test type: Other — Mixed-effects model; p < 0.01, Mixed Models Analysis — Main effect of time; F(1, 26) = 33.29
Statistical Analysis 3: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; UEMS; Test type: Other — Mixed-effects model; p = 0.04, Mixed Models Analysis — Treatment group by time interaction effects; F(1,26) = 4.58
Statistical Analysis 4: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; UEMS; Test type: Other — Mixed-effects model; p < 0.01, Mixed Models Analysis — Main effect of time; F(1, 26) = 15.34
Statistical Analysis 5: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; TMS; Test type: Other — Mixed-effects model; p < 0.01, Mixed Models Analysis — Treatment group by time interaction effects; F(1,26) = 8.06
Statistical Analysis 6: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Test type: Other — TMS; p < 0.01, Mixed Models Analysis — Main effect of time; F(1,26) = 38.91
Statistical Analysis 7: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; TLTS; Test type: Other — Mixed-effects model; p = 0.02, Mixed Models Analysis — Treatment group by time interaction effects; F(1,21.7) = 6.23
Statistical Analysis 8: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; TLTS; Test type: Other — Mixed-effects model; p = 0.05, Mixed Models Analysis — Main effect of time; F(1 26)=4.14

3. Secondary Outcome: Change in International Spinal Cord Injury Basic Pain Data Set (ISCIBPDS) 2.0
Description: Change in International Spinal Cord Injury Basic Pain Data Set (ISCIBPDS) 2.0 contains critical questions about clinically relevant information concerning SCI-related pain during the last 7 days, including pain intensity, the influence of pain on daily activities, mood, and sleep between admission and discharge. Full scale from 0-10, higher score indicates more pain.
Time Frame: Baseline and at discharge from acute inpatient rehabilitation (average 2-3 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exoskeletal-assisted Walking Training Group | Standard of Care Group
Number analyzed (Participants) | 16 | 12
score on a scale
  Average worst pain intensity | 4.9 (3.6) | 3.7 (4.4)
  Worst pain interference with day-to-day activities | 2.4 (3.9) | 2.0 (5.3)
  Worst pain interference with overall mood | 3.6 (4.7) | 2.7 (6.2)
  Worst pain interference with sleep | 3.5 (4.0) | 3.4 (5.5)
Statistical Analysis 1: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Average worst pain intensity; Test type: Other — Mixed-effects model; p = 0.485, Mixed Models Analysis — Treatment group-by-time interaction effect; F(1, 21) = 0.51
Statistical Analysis 2: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Average worst pain intensity; Test type: Other — Mixed-effects model; p = 0.000, Mixed Models Analysis — Main effect of time; F(1, 21) = 26.71
Statistical Analysis 3: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Worst pain interference with day-to-day activities; Test type: Other — Mixed-effects model; p = 0.832, Mixed Models Analysis — Treatment group-by-time interaction effect; F(1, 21) = 0.05
Statistical Analysis 4: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Worst pain interference with day-to-day activities; Test type: Other — Mixed-effects model; p = 0.033, Mixed Models Analysis — Main effect of time; F(1, 21) = 5.21
Statistical Analysis 5: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Worst pain interference with overall mood; Test type: Other — Mixed-effects model; p = 0.692, Mixed Models Analysis — Treatment group-by-time interaction effect; F(1, 42) = 0.16
Statistical Analysis 6: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Worst pain interference with overall mood; Test type: Other — Mixed-effects model; p = 0.005, Mixed Models Analysis — Main effect of time; F(1, 42) = 8.65
Statistical Analysis 7: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Worst pain interfered with sleep; Test type: Other — Mixed-effects model; p = 0.946, Mixed Models Analysis — Treatment group-by-time interaction effect; F(1,21) = 0.01
Statistical Analysis 8: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Worst pain interference with sleep; Test type: Other — Mixed-effects model; p = 0.0002, Mixed Models Analysis — Main effect of time; F(1,21) = 11.94

4. Secondary Outcome: Number of Participants With Neuropathic Pain
Description: Number of participants with neuropathic pain as measured by the Spinal Cord Injury Pain Instrument (SCIPI).
  Spinal Cord Injury Pain Instrument (SCIPI) is a tool used to classify pain after SCI using 4 questions. It can be easily used by clinicians in every clinical setting to identify the pain classifications, including neuropathic, nociceptive, neither or unknown. Full scale from 0 to 4, a score of 1 or more than 1 indicates probable neuropathic pain.
Time Frame: Baseline and discharge from acute inpatient rehabilitation (average 2-3 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Exoskeletal-assisted Walking Training Group | Standard of Care Group
Number analyzed (Participants) | 12 | 11
Participants
  Baseline | 3 | 4
  discharge from acute inpatient rehabilitation (average 2-3 weeks) | 1 | 1
Statistical Analysis 1: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; Baseline; Test type: Superiority; p = 0.554, Chi-squared; X^2 (1, N = 23) = 0.35
Statistical Analysis 2: Comparison: Exoskeletal-assisted Walking Training Group vs Standard of Care Group; discharge from acute inpatient rehabilitation (average 2-3 weeks); Test type: Superiority; p = 0.949, Chi-squared; X^2 (1, N = 23) = 0.004

ADVERSE EVENTS:
Time Frame: Average 2-3 weeks
Arm/Group | Exoskeletal-assisted Walking Training Group | Standard of Care Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 5/16 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exoskeletal-assisted Walking Training Group (N=16) | Standard of Care Group (N=12)
right trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
severe Orthostatic Hypotension (Nervous system disorders) | 1 | 0
left-hand numbness (Nervous system disorders) | 1 | 0
device malfunction-related events (Product Issues) | 2 | 0

LIMITATIONS AND CAVEATS:
Small sample size and potential selection bias due to the lack of a prospectively randomized comparison group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT04221373/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT04221373/ICF_001.pdf